CLINICAL TRIAL: NCT06861049
Title: The Effect of Psychobiotic Use on Mental Health, Quality of Life, Anthropometric and Biochemical Outcomes in Obese Women on a Weight-loss Diet
Brief Title: Psychobiotics and Mental Health in Obese Women on a Weight-Loss Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Rabia Melda Karaağaç, Principal Investigator, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IMU-BES-RMK-01
Record Dates: First submitted 2025-02-27; First posted 2025-03-06 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Obesity; Mental Health; Probiotic
MeSH Terms: conditions — Obesity; Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Psychobiotic Group (Experimental): Participants will receive a psychobiotic supplement along with a weight-loss diet.
  Interventions: Dietary Supplement: Psychobiotic Supplement
- Placebo Group (Placebo Comparator): Participants will receive a placebo supplement along with a weight-loss diet.
  Interventions: Dietary Supplement: Placebo Supplement

INTERVENTIONS:
Dietary Supplement: Psychobiotic Supplement — Lactobacillus helveticus R0052 Bifidobacterium bifidum R0071 Bifidobacterium longum R0175
  Arms: Psychobiotic Group
Dietary Supplement: Placebo Supplement — Maltodextrin
  Arms: Placebo Group

SUMMARY:
The aim of this study was to evaluate the effect of psychobiotic supplementation containing Lactobacillus helveticus R0052, Bifidobacterium bifidum R0071 and Bifidobacterium longum R0175 strains on mental health, quality of life, anthropometric measurements and some biochemical parameters in obese women. In the randomized double-blind placebo-controlled study, 28 obese female participants (14 psychobiotic, 14 placebo) will be given psychobiotic supplement/placebo together with a weight loss diet once a day every day for 4 weeks. Before and after the intervention, anthropometric measurements, blood samples and 24-hour retrospective 3-day food consumption records of the participants will be taken. In addition, the Depression Anxiety Stress Scale (DASS-21) will be administered to measure mental health, the SF-36 Quality of Life Scale to determine quality of life, and the International Physical Activity Questionnaire (IPAQ) to determine physical activity levels. Psychobiotics, which have entered our lives in recent years, have many beneficial effects on mental health through gut microbiota. However, while the effects of psychobiotics on mental health have been studied, their effects on obesity have not been investigated much. This study is unique in that it is the first study to investigate the effect of psychobiotic use on mental health in obese individuals. However, obesity is known to be an inflammatory disease and there is no study in the literature that includes the systemic immune inflammation index (SII) as a biomarker. SII is effective in evaluating the inflammatory and immune response in the body and determining prognosis; it adds value to clinical practice with early diagnosis of diseases, treatment follow-up and a wide range of uses.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged ≥ 18-65 years
* BMI ≥30 kg/m2
* Willingness to volunteer
* Able to give written consent

Exclusion Criteria:

* Co-administration of probiotics. However, subjects will be eligible to participate after a four (4) week washout period.
* Pregnant or planning to become pregnant within the next two (2) months.
* Positive pregnancy test in women of childbearing potential.
* Use of antibiotic medication (e.g. neomycin, rifaximin) within the last 1 month. If this is the case, the participant will be eligible to participate four (4) weeks after completion of antibiotic treatment (washout period).
* Individuals with physician-diagnosed psychiatric and neurological conditions.
* Individuals with irritable bowel syndrome or gastrointestinal disorders.
* People with immune disorders or possible immunodeficiency states (e.g. due to surgery).
* Use of anti-inflammatory drugs
* Use of corticosteroids
* People who are allergic to milk, corn starch or soya.
* Foreign nationality.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 40 (Actual)
Dates: Start 2025-02-13 (Actual); Primary Completion 2025-07-03 (Actual); Study Completion 2025-07-03 (Actual)

PRIMARY OUTCOMES:
Changes in Body Weight (kg) from Baseline to Week 4 | Baseline and Week 4
Changes in Body Mass Index (BMI) from Baseline to Week 4 | Baseline and Week 4
  Body Mass Index (BMI) will be calculated as weight (kg) / height (m²). Higher BMI values indicate higher body fatness.

SECONDARY OUTCOMES:
Changes in mental health status with DASS-21 from Baseline to Week 4 | Baseline and Week 4
  Depression, Anxiety, and Stress Scale-21 (DASS-21). Scores range from 0 to 63 for each subscale, with higher scores indicating worse mental health status.
Changes in Quality of Life with SF-36 from Baseline to Week 4 | Baseline and Week 4
  Short Form-36 Health Survey (SF-36). Scores range from 0 to 100, with higher scores indicating better quality of life.
Changes in C-Reactive Protein (CRP) Levels from Baseline to Week 4 | Baseline and Week 4
  C-reactive protein (CRP) measured in mg/L. Higher values indicate greater inflammation.
Changes in Interleukin-6 (IL-6) Levels from Baseline to Week 4 | Baseline and Week 4
  Interleukin-6 (IL-6) measured in pg/mL. Higher values indicate greater inflammation.
Changes in Systemic Immune-Inflammation Index (SII) from Baseline to Week 4 | Baseline and Week 4
  SII calculated as (Platelets × Neutrophils) / Lymphocytes. Higher scores indicate higher systemic inflammation.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No